CLINICAL TRIAL: NCT00685243
Title: Treatment of Surgical Scars With Fractional Photothemolysis Versus Pulse Dye Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: American Academy of Cosmetic Surgery (Other)
Responsible Party: Principal Investigator, David M. Ozog, Chair, Department of Dermatology, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB4812
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Post Surgical Scars
Keywords: Fraxel; Pulsed dye laser; Surgical scars
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fraxel (Active Comparator): Fraxel laser treatment
  Interventions: Procedure: Laser treatment
- PDL (Active Comparator): Pulsed dye laser treatment
  Interventions: Procedure: Laser treatment

INTERVENTIONS:
Procedure: Laser treatment — Fraxel and pulsed dye laser
  Other Names: -Fraxel SR Laser (Reliant Technologies, Inc.); -V-Beam Pulse Dye laser (Candela Corporation)

SUMMARY:
1. Evaluate the efficacy of the Fraxel SR laser to improve the cosmetic appearance of surgical scars, both in terms of pigmentary and textural changes.
2. Evaluate the efficacy of the V-Beam Pulse Dye laser, a standard non-ablative laser which is utilized for the treatment of the erythematous and telangiectasia component of surgical scars.
3. Comparison of the outcome of the half of the surgical scar treated with Fraxel SR laser versus the outcome of the contralateral half of the surgical scar which will be treated with the V-Beam Pulse Dye Laser.

DETAILED DESCRIPTION:
RATIONALE FOR THE PROJECT

Surgical scars are a challenging condition to treat. The aesthetic outcome of surgical scars is of great importance to patients and physicians after reconstructive surgery. The current approaches for the treatment of surgical scars range from non-invasive approaches to aggressive treatments with re-excision or ablative resurfacing lasers. Fractional photothemolysis is a new technology whereby only microthermal zones of injury to the skin are created which triggers the wound healing response, leading to skin repair mechanisms to improve the appearance and textural changes associated with surgical scars.

Fractional photothemolysis (Fraxel SR laser, Reliant technologies, Inc) is a new technology whereby only microthermal zones of injury to the skin are created which triggers the wound healing response, leading to skin repair mechanisms to improve the appearance and textural changes associated with surgical scars. Fractionated resurfacing, with its significant proven efficacy in improving textural and pigmenatary abnormalities with a benign side effect profile, represents a promising novel treatment for surgical scars.

Aim:

Comparison of the outcome of the half of the surgical scar treated with Fraxel SR (Reliant Technologies, Inc.) laser versus the outcome of the contralateral half of the surgical scar which will be treated with the V-Beam Pulse Dye Laser

SIGNIFICANCE:

The cosmetic outcome of surgical scars is of paramount importance to surgeons and patients treated with both cosmetic and reconstructive surgery. It is impossible for surgeons to predict the wound healing properties of individual patients and particular anatomic sites and thus, there is little certainty that can be offered to patients about the cosmetic outcome of their surgical scars.

SUBJECTS IN THE PROJECT:

Inclusion Criteria:

For inclusion, the subject must:

1. Be at least 18 years old;
2. Be otherwise healthy;
3. Be treated by Dr. Kouba for a skin cancer surgery or plastic surgery procedure
4. Agree to attend up 6 sessions post Mohs surgery (2-4 laser treatment sessions and 2 follow-up visits post-laser)
5. Be able to understand the requirements of the study, the risks involved, and be able to sign the informed consent form;
6. Agree to follow and undergo all study-related procedures.

Exclusion criteria:

A. Patients who do not meet the criteria above and/or who fail to follow their post-operative instructions or make both of their post-operative clinic appointments.

B. The control for this study will be the side of the scar treated with the V-Beam Pulse Dye Laser

C. We will be speaking to patients at Henry Ford Dermatology regarding participation in our study. We will ensure that all patients understand the voluntary nature of their participation in the study. They will sign informed consent. In addition, we will be asking patients to give us their assessment of which side of their surgical wound had better improvement, the side treated with Fraxel laser versus the side treated with V-Beam Pulse Dye Laser.

PROJECT DESIGN AND PROCOTOL:

1. A comparison trial of surgical scars treated with Fraxel SR Laser (Reliant Technologies, Inc.) versus V-Beam Pulse Dye Laser (Candela Corporation) in 15 patients who underwent Mohs surgery and resultant cosmetic surgical reconstruction at Henry Ford Health System Department of Dermatology.
2. At a minimum of 2 months post surgical reconstruction, patients will be eligible for inclusion in this research study. During each 2 weeks of the study, one side of the surgical scar will be treated with Fraxel SR (Reliant Technologies, Inc.) and the other half will be treated with the V-Beam Pulse Dye Laser (Candela Corporation) for aesthetic improvement of the scar

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years old;
2. Be otherwise healthy;
3. Be treated by Dr. Kouba for a skin cancer surgery or plastic surgery procedure
4. Agree to attend up 6 sessions post Mohs surgery (2-4 laser treatment sessions and 2 follow-up visits post-laser)
5. Be able to understand the requirements of the study, the risks involved, and be able to sign the informed consent form;
6. Agree to follow and undergo all study-related procedures.

Exclusion Criteria:

1. Patients who do not meet the criteria above and/or who fail to follow their post-operative instructions or make both of their post-operative clinic appointments.
2. The control for this study will be the side of the scar treated with the V-Beam Pulse Dye Laser
3. We will be speaking to patients at Henry Ford Dermatology regarding participation in our study. We will ensure that all patients understand the voluntary nature of their participation in the study. They will sign informed consent. In addition, we will be asking patients to give us their assessment of which side of their surgical wound had better improvement, the side treated with Fraxel laser versus the side treated with V-Beam Pulse Dye Laser.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Overall cosmetic appearance, relative to adjacent skin and side effects. | 6 months

SECONDARY OUTCOMES:
skin matches surrounding skin, no scar formation visible, skin pigmentation and/or texture of scarred region is markedly different from surrounding skin). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Kouba, MD, PhD, Principal Investigator — Department of Dermatology, Henry Ford Health System
Locations (1):
- Department of Dermatology, Henry Ford Medical Center, 6530 Farmington Rd, West Bloomfield, Michigan, United States

REFERENCES:
- [Background] Alster TS. Improvement of erythematous and hypertrophic scars by the 585-nm flashlamp-pumped pulsed dye laser. Ann Plast Surg. 1994 Feb;32(2):186-90. doi: 10.1097/00000637-199402000-00015. PMID 8192370
- [Background] Behroozan DS, Goldberg LH, Dai T, Geronemus RG, Friedman PM. Fractional photothermolysis for the treatment of surgical scars: a case report. J Cosmet Laser Ther. 2006 Apr;8(1):35-8. doi: 10.1080/14764170600607251. PMID 16581684